CLINICAL TRIAL: NCT00298545
Title: High vs. Low Calcium Intake in the Presence of High Vitamin D: Effect on Gene Expression in the Colon
Brief Title: Effect of Vitamin D and Calcium on Genes in the Colon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: RUH IRB # PHO-0554
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Colorectal Polyps; Colorectal Adenoma; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Calcitriol; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo and Calcitriol (Placebo Comparator): placebo tablets together with an oral tablet of 1, 25 dihydroxy vitamin D3 (Calcitriol)
  Interventions: Drug: placebo and Calcitriol
- 2 (Active Comparator): calcium together with an oral tablet of 1, 25 dihydroxy vitamin D3 (Calcitriol)
  Interventions: Drug: Calcium and Calcitriol

INTERVENTIONS:
Drug: placebo and Calcitriol — Placebo tablets twice daily together with an oral tablet of 1, 25 dihydroxy vitamin D3 (Calcitriol)
  Arms: placebo and Calcitriol
Drug: Calcium and Calcitriol — Calcium twice daily together with an oral tablet of 1, 25 dihydroxy vitamin D3 (Calcitriol)
  Arms: 2

SUMMARY:
The researchers are involved in a research program to understand how vitamin D and calcium in the diet or as supplements may lower the risk of colorectal polyps and cancer. To that end, the researchers are conducting a study of vitamin D supplementation in which volunteer subjects are provided a Western style diet for 2 separate 4 week periods at the Rockefeller University Hospital. During one of these 4 week inpatient periods, subjects receive calcium supplements and during the other 4 week inpatient period they receive a placebo tablet. The researchers determine changes within the colon as a result of supplementing the vitamin D in the presence of high and low calcium. A more detailed description of the study is provided below.

DETAILED DESCRIPTION:
Study subjects participate for about 3 months. During this time, there is one outpatient visit, a 4 week inpatient period, a 4 week outpatient period known as a wash out period and finally another 4 week inpatient period. During the inpatient periods, the Rockefeller University Hospital (RUH) becomes your home. The subject must sleep here every night and consume all the food provided. During the screening visit, blood and urine samples will be taken and an EKG (electrocardiogram) and a complete physical exam will be done. After enrollment into the study, the first 4 week inpatient period begins. You may continue to go to work or do other activities as long as you eat the diet provided and sleep at the Rockefeller University Hospital. You must eat everything that we give you and you may not substitute or supplement the diet in any way. During each 4 week stay at the Rockefeller University Hospital, there will be three flexible sigmoidoscopies done and biopsies taken of the mucosal lining of the colorectum. This procedure is painless and takes about 5 minutes. In addition, blood samples will be taken every few days for follow-up and research, and two 24 hour urine samples will be done on separate days during the hospitalization. Vital signs are measured every day and your weight will be measured three times per week. During the four week wash out period, the subject will return to their home, go about their normal activities and consume their normal diet. The subject will return to the Rockefeller University Hospital for the second 4 week inpatient period. The procedures and laboratory tests are the same during the second inpatient period. The study concludes with the subjects' discharge from the RUH.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers with a history of pre-cancerous colorectal polyps and/or have a family history of pre-cancerous polyps or colon cancer
2. Not taking any medications known to affect either calcium metabolism or colon function
3. Between the ages of 48 and 72 years old
4. Have had pre-cancerous colorectal polyps or have first or second degree relatives with colorectal cancer and are therefore at increased risk for the disease

Exclusion Criteria:

1. Personal history of cancer other than non-melanoma skin cancer
2. Diseases of the bowel such as intestinal malabsorption or inflammatory bowel disease
3. Prior gastrointestinal surgery including gastrectomy, small or large bowel resections. (If one has had an appendectomy or surgery of the esophagus, he/she is still eligible.)
4. Any excessive bleeding or clotting disorders
5. Taking blood thinners
6. Abnormalities of or conditions predisposing one to abnormalities of calcium metabolism. (This includes untreated hyperparathyroidism [increase in parathyroid function] and history of milk-alkali syndrome, a type of calcium metabolism disease.)
7. Untreated hyperthyroidism (increase in thyroid function)
8. Regularly take greater than 660 mg of aspirin per day. This is greater than two tablets of 325 mg regular strength aspirin or greater than one tablet of 500 mg of extra strength aspirin per day. (If one has been taking aspirin for heart or blood vessel protection regularly for at least one month before his/her first screening visit, he/she will remain on the same amount of medicine throughout the study. The following amounts are acceptable:

   * Aspirin 1 to 2 regular tablets (325 mg) per day, or
   * Baby aspirin 1 tablet (81 mg) per day
9. Regularly take daily dosages of nonsteroidal anti-inflammatory agents (NSAIDs) within the last 3 months. (One example of an NSAID is ibuprofen.)
10. Taking greater than 1200 mg of dietary calcium daily
11. Taking medications called sterol-binding resins, such as cholestyramine (Questran®), which is for the treatment of high blood cholesterol
12. Taking other investigational drugs or multiple other medications that might, in the opinion of the investigator, affect the study measurements.
13. Other serious illness(es) that are anticipated to limit life expectancy to less than 6 months
14. Elevated blood pressure greater than 160/100 mmHg
15. HIV positive
16. Pregnant or nursing
17. A history of kidney stones
18. Liver disease and/or kidney disease
19. Diabetes mellitus
20. High "bad" cholesterol level, low density lipoprotein (LDL) greater than 175 mg/dl or triglyceride levels greater than 600 mg/dl
21. Known history of coronary artery disease
22. EKG (electrocardiogram is a record of the electrical activity of the heart) changes consistent with a past heart attack (myocardial infraction)
23. Currently taking:

    * Antidiabetic medication
    * Hormone replacement therapies, oral, injected or implanted contraceptives. (Thyroid hormone replacement is allowed as long as one's thyroid test is normal.)
    * Vitamin, mineral, fish oil, and herbal supplementation and weight control medication must be stopped at least 1 month prior to enrolling in the study.

Ages: 48 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Gene expression related to proliferation, apoptosis, and differentiation of human rectal mucosal cells | end of study

SECONDARY OUTCOMES:
Expression of additional genes involved in the cell properties noted above | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Holt, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Protiva P, Pendyala S, Nelson C, Augenlicht LH, Lipkin M, Holt PR. Calcium and 1,25-dihydroxyvitamin D3 modulate genes of immune and inflammatory pathways in the human colon: a human crossover trial. Am J Clin Nutr. 2016 May;103(5):1224-31. doi: 10.3945/ajcn.114.105304. Epub 2016 Mar 23. PMID 27009752